#### **Short Title:**

# Statistical Analysis Plan CLL949-C018 / NCT04207749

**Full Title:** 

Statistical Analysis Plan CLL949-C018

| Protocol Title: | Clinical Evaluation of a Daily Wear Silicone Hydrogel Lens |
|---|---|
| Project Number: | |
| Reference Number: | |
| Protocol TDOC Number: | TDOC-0056860 |
| Author: | |
| Approvals: | See last page for electronic approvals. |
| Job Notes: | |

This is the first revision (Version 2.0) of the Statistical Analysis Plan for this study. This version of the Statistical Analysis Plan is based on Version 2.0 of the study protocol.

Document ID: V-CLN-0002343 Page 2 of 23

Status: Approved, Version: 2.0 Approved Date: 05 Jan 2021

# **Executive Summary:**

| Zaccutive Summury. |
|---|
| Key Objectives: |
| The primary effectiveness objective is to demonstrate noninferiority of soft contact lenses compared to BIOFINITY® soft contact lenses (Biofinity), in contact lens corrected distance visual acuity (CLCDVA) at Week 1 Follow-up. |
| The secondary effectiveness objective is to demonstrate noninferiority of compared to Biofinity in the percentage of subjects achieving CLCDVA 20/20 or better, in each eye, at Week 1 Follow-up. |

# **Table of Contents**

| Statistic | al Analysis Plan CLL949-C018 | 1 |
|---|---|---|
| Table of | Contents | 3 |
| List of T | Tables | 4 |
| 1 | Study Objectives and Design | 5 |
| 1.1 | Study Objectives | 5 |
| 1.2 | Study Description | |
| 1.3 | Randomization | 6 |
| 1.4 | Masking | 6 |
| 2 | Analysis Sets | 7 |
| 2.1 | Safety Analysis Set | 7 |
| 2.2 | Full Analysis Set | |
| 2.3 | Per Protocol Analysis Set | 7 |
| 3 | Subject Characteristics and Study Conduct Summaries | 8 |
| 4 | Effectiveness Analysis Strategy | 8 |
| 4.1 | Effectiveness Endpoints | 9 |
| 4.2 | Effectiveness Hypotheses | 10 |
| 4.3 | Statistical Methods for Effectiveness Analyses | 10 |
| 4.3.1<br>4.3.2 | Primary Effectiveness Analyses | |
| 5 | Safety Analysis Strategy | 12 |
| 5.1 | Safety Endpoints | |
| 5.2 | Safety Hypotheses | |
| 5.3 | Statistical Methods for Safety Analyses | |
| <ul><li>5.3.1</li><li>5.3.2</li></ul> | Adverse Events | |

Page 4 of 23

| 5.3.3 | Device Deficiencies | 15 |
|---|---|---|
| 8 | Other Reporting Considerations and Analysis Strategies | 1 <i>6</i> |
| 9 | References | 17 |
| 11 | Appendix | 20 |
| | List of Tables | |
| Table 1 | -1 Study Description Summary | 5 |
| Table 8 | -1 Analysis Windows | 16 |
| Table 1 | 1-1 Schedule of Study Procedures and Assessments | 20 |

# 1 Study Objectives and Design

To address the primary and secondary effectiveness objectives, data from a pre-determined subset of subjects from CLL949-C009 will be combined with data from the current study, and all planned analyses will be performed on the combined set of data.

## 1.1 Study Objectives

#### PRIMARY OBJECTIVE

The primary effectiveness objective is to demonstrate noninferiority compared to Biofinity in mean CLCDVA at Week 1 Follow-up.

#### **SECONDARY OBJECTIVE**

The secondary effectiveness objective is to demonstrate noninferiority compared to Biofinity in the percentage of subjects achieving CLCDVA 20/20 or better, in each eye, at Week 1 Follow-up.

## 1.2 Study Description

Key components of the study are summarized in Table 1-1.

**Table 1-1 Study Description Summary** 

| Study Design | Prospective, multi-center, randomized,, controlled, |
|---|---|
| | double-masked, parallel-group |
| Study Population | Volunteer subjects aged 18 or over who are adapted daily wear |
| | frequent replacement soft contact lens wearers, excluding |
| | Biofinity habitual wearers, have at least 3 months of soft contact |
| | lens wearing experience, and who wear their habitual lenses at |
| | least 5 days per week and at least 8 hours per day. |
| | reast 5 days per week and at reast 6 nours per day. |

| | Target to complete: 192 subjects (128:64; Test:Control) Planned: ~252 subjects enrolled, ~228 subjects randomized (152:76; Test:Control) |
|---|---|
| Number of Sites | ~14-17 (US) |
| Test Product | soft contact lenses |
| Control Product | CooperVision® BIOFINITY® (comfilcon A) soft contact lenses |
| | (Biofinity) |
| Duration of Treatment | Approximately 3 months |
| Visits | Visit 1: Screening/Baseline/Dispense (Day 1) |
| | Visit 2: Week 1 Follow-up |
| | Visit 3: Month 1 Follow-up |
| | Visit 4: Month 3 Follow-up/Exit |

## 1.3 Randomization

A member of the Randomization Programming group at Alcon who is not part of the study team will generate the randomized allocation schedule(s) for study lens assignment.

| Subjects will be randomized in a 2:1 ratio to receive either lenses, respectively. | or Biofinity contact |
|---|---|

# 1.4 Masking

This study is double-masked.



## 2 Analysis Sets

Data from a subset of subjects in the CLL949-C009 study will be combined with data from this study. This combined set will serve as the basis for all analyses for the primary and secondary effectiveness objectives. Subjects in CLL949-C009 will be included in the combined set only if they satisfy the following criterion:

 Best corrected visual acuity (BCVA) of 20/20 or better in each eye at the Screening / Baseline / Dispense Visit

## 2.1 Safety Analysis Set

| Safety analyses will be conducted using the safety analysis set on a treatment-emergent basis |
|---|
| As such, the safety analysis set will include all subjects/eyes exposed to any study lenses |
| evaluated in this study. |
| For treatment-emergent |
| safety analyses, subjects/eyes will be categorized under the actual study lenses exposed. |

# 2.2 Full Analysis Set

The full analysis set (FAS) is the set of all randomized subjects who are exposed to any study lenses evaluated in this study, and who have at least one post-baseline (post-Dispense) CLCDVA.

# 2.3 Per Protocol Analysis Set

The per protocol (PP) analysis set is a subset of FAS and excludes all data/subjects that have met any of the critical deviation or evaluability criteria identified in the Deviations and Evaluability Plan (DEP).

# 3 Subject Characteristics and Study Conduct Summaries

Demographic information (age, sex, ethnicity, and race), recent lens-wearing experience (wear modality, wear success), and habitual lens information will be presented by lens group and overall for the safety, full, and per protocol analysis sets.

Baseline data will also be summarized by lens group and overall on the safety, full and per protocol analysis sets.



All data obtained in evaluable subjects/eyes will be included in the analysis. No imputation for missing values will be carried out for the effectiveness analyses.

For all planned inferential analyses, alternative models/methods may be considered if convergence cannot be achieved.

# 4.1 Effectiveness Endpoints

### **Primary Endpoint**

The primary endpoint is the mean CLCDVA at Week 1 Follow-up. The corresponding assessment is collected with study lenses, in Snellen, for each eye. Conversion will be made to the logMAR scale.

## **Secondary Endpoint**

The secondary endpoint is the percentage (proportion) of subjects with CLCDVA of 20/20 or better, measured monocularly, in both OD and OS at Week 1 Follow-up.





# 4.2 Effectiveness Hypotheses

#### **Primary Effectiveness**

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.10 (in logMAR scale) for noninferiority:

H<sub>0</sub>: 
$$\mu_{(T)} - \mu_{(C)} \ge 0.10$$
  
H<sub>a</sub>:  $\mu_{(T)} - \mu_{(C)} < 0.10$ 

where  $\mu_{(T)}$  and  $\mu_{(C)}$  denote the Week 1 Follow-up mean CLCDVA for Mercury and Biofinity, respectively, on the logMAR scale.

#### **Secondary Effectiveness**

The null and alternative hypotheses are formulated in terms of the predefined margin of 0.10 (10%) for noninferiority.

$$H_0: P_{(T)} - P_{(C)} \le -0.10$$
  
 $H_a: P_{(T)} - P_{(C)} > -0.10$ 

where  $P_{(T)}$  and  $P_{(C)}$  denote the proportion of subjects attaining at least 20/20 in CLCDVA at Week 1 Follow-up in each eye (OD and OS) for Mercury and Biofinity, respectively.

# 4.3 Statistical Methods for Effectiveness Analyses

# **4.3.1** Primary Effectiveness Analyses

A mixed effects repeated measures model will be utilized to test these hypotheses.

Lens difference (Mercury minus Biofinity) and the

corresponding two-sided 95% CI will be computed for Week 1 Follow-up. Noninferiority in CLCDVA will be declared if the upper confidence limit is less than 0.10.





Biofinity), noninferiority in proportion of subjects achieving 20/20 or better in CLCDVA in both eyes will be declared if the lower confidence limit is greater than -0.10.





## 5.1 Safety Endpoints

The safety endpoints are:

- Adverse Events (AEs)
- Biomicroscopy Findings



• Device Deficiencies

# 5.2 Safety Hypotheses

There are no safety hypotheses planned in this study. The focus of the safety analysis will be a comprehensive descriptive assessment of safety endpoints listed in Section 5.1.

# 5.3 Statistical Methods for Safety Analyses

#### 5.3.1 Adverse Events

The applicable definition of an AE is in the study protocol. All AEs occurring from when a subject signs informed consent to when a subject exits the study will be accounted for in the reporting. Analysis and presentation of pre-treatment AEs will be separated from treatment-emergent AEs occurring during the study period. A pre-treatment AE is an event that occurs after signing informed consent but prior to exposure to the study lens (not including trial fitting lenses). The period for treatment-emergent AE analysis starts from exposure to study lens until the subject completes or is discontinued from the study.

Descriptive summaries (counts and percentages) for ocular and nonocular AEs will be presented by Medical Dictionary for Regulatory Activities (MedDRA) Preferred Terms (PT). Serious AEs and significant non-serious ocular AEs will be noted. Additionally, relationship to lens will be identified in all AE tables. Unit of presentation for ocular AEs will be eye and nonocular AEs will be subject.

Individual subject listings will be provided for both pre-treatment and treatment-emergent AEs, where any AE leading to study discontinuation will be indicated.

## 5.3.2 Biomicroscopy Findings/Slit Lamp Examination

Biomicroscopy assessment will be performed at all study visits, including Screening/Baseline/Dispense, Week 1 Follow-up, Month 1 Follow-up, Month 3 Follow-up and unscheduled visits. The reporting unit for each biomicroscopy finding will be eye.

# 5.3.3 Device Deficiencies

A frequency table showing counts for each treatment-emergent Device Deficiency category will be presented. In addition, listings for treatment-emergent and pre-treatment device deficiencies will be provided.

| _ |
|---|
| ı |
| - |
| • |



Document ID: V-CLN-0002343

Status: Approved, Version: 2.0 Approved Date: 05 Jan 2021



# 9 References

1. ISO 11980:2012 Ophthalmic optics - Contact lenses and contact lens care products - Guidance for clinical investigations





# 11 Appendix

**Table 11-1 Schedule of Study Procedures and Assessments** 

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense Day 1 | Visit 2 Week 1 Follow-up Day 7 | Visit 3 Month 1 Follow-up Day 30 | Visit 4 Month 3 Follow-up/ Exit Day 95 | Early<br>Exit | USV |
|---|---|---|---|---|---|---|
| Informed Consent | ✓ | - | - | - | - | - |
| Demographics | ✓ | - | - | - | - | - |
| Medical History | ✓ | ✓ | ✓ | ✓ | ✓ | <b>(√)</b> |
| Concomitant<br>Medications | <b>√</b> | ✓ | <b>√</b> | <b>√</b> | <b>✓</b> | (✔) |
| Inclusion/ Exclusion | ✓ | - | - | - | - | - |
| Habitual lens information (brand / manufacturer, modality, power, wear success, habitual lens care brand) | <b>√</b> | - | - | - | - | - |
| VA w/ habitual<br>correction (OD,OS<br>Snellen distance) | ✓ | - | - | <b>√</b> | <b>✓</b> | <b>(√)</b> |
| | - | ı | | • | | |
| | | | F | | | |
| | - | C | _ | - | • | |
| Biomicroscopy <sup>2</sup> | ✓ | ✓ | ✓ | ✓ | ✓ | <b>(√)</b> |
| | | I | | | | |

| Procedure/ Assessment | Visit 1 Screening/ Baseline/ Dispense Day 1 | Visit 2 Week 1 Follow-up Day 7 | Visit 3 Month 1 Follow-up Day 30 | Visit 4 Month 3 Follow-up/ Exit Day 95 | Early<br>Exit | USV |
|---|---|---|---|---|---|---|
| | | 1 | 1 | 1 | 1 | - |
| Randomize | ✓ | - | - | - | - | - |
| IP Dispense | ✓ | ✓ | (✓) | - | - | (✔) |
| VA w/ study lenses<br>(OD, OS Snellen<br>distance) | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>√</b> | <b>(√)</b> |

| | Visit 1 | Visit 2 | Visit 3 | Visit 4 | | |
|---|---|---|---|---|---|---|
| Procedure/ Assessment | Screening/<br>Baseline/<br>Dispense | Week 1<br>Follow-up | Month 1<br>Follow-up | Month 3<br>Follow-up/<br>Exit | Early<br>Exit | USV |
| | Day 1 | Day 7 | Day 30 | Day 95 | | |

| AEs | ✓ | ✓ | ✓ | ✓ | ✓ | <b>(√)</b> |
|---------------------|-----|-----|-----|---|---|------------|
| Device deficiencies | ✓ | ✓ | ✓ | ✓ | ✓ | (✓) |
| Exit Form | (✓) | (✓) | (✓) | ✓ | ✓ | (✓) |



Signature Page for V-CLN-0002343 v2.0

